CLINICAL TRIAL: NCT00498381
Title: The Induction of IL-6 by NF-kB in PBMC in OSA
Acronym: OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9361701235
Record Dates: First submitted 2007-07-08; First posted 2007-07-10 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2005-02

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CPAP

SUMMARY:
Aim of study:

1. To compare the level of IL-6 mRNA expression in peripheral blood monocytes between normal subjects and patients with OSAS
2. To compare the activation of NF-B in peripheral blood monocytes between control subjects and patients with OSAS; Check the correlation between level of L-6 mRNA expression and activation of NF-kB
3. To determine the effect of CPAP on the activation of NF-kB and IL-6 in peripheral blood monocytes in patients with moderate -severe OSAS

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) has emerged in recent years as an important risk factor for cardiovascular morbidity. The mechanisms responsible for developments of cardiovascular sequelae in patients with OSA include hypoxia, hypercapnia, exaggerated negative intrathoracic pressure and bursts of sympathetic activity provoking surges in blood pressure and heart rate. Meanwhile, increase of inflammatory mediators, which included C-reactive protein (CRP), oxidative stress, adhesion molecules, vascular endothelial growth factor (VEGF) and proinflammatory cytokines (interleukin (IL) -1, IL-2, IL-6, IL-8, IL-10 and tumor necrotic factor- (TNF-)), also involve in the development of cardiovascular disease in patients with OSAS.

According to our preliminary study, serum levels of IL-6 and CRP were higher in patients with OSAS than control subjects and levels of both IL-6 and CRP were highly correlated with the lowest pulse oxygen saturation. Hypoxia triggered the production of IL-6 through the induction of NFB, which was demonstrated in ischemic heart disease and pancreatitis. However, this mechanism has not been prooved in OSAS.

Therefore, we conduct this study to prove our hypothesis (1) The mRNA expression of IL-6 in peripheral blood monocytes was significantly higher in patients with OSAS than control subjects (2) The activation of NF-k B in peripheral blood monocytes was more significant in patients with OSAS than control subjects, and the level of NF- kB activation is associated with the level of IL-6 mRNA expression (3) CPAP therapy could lower both the activation of NF-kB and IL-6 mRNA expression in patients with moderate-severe OSAS.

ELIGIBILITY:
Inclusion Criteria:

* severe obstructive sleep apnea (AHI>=30 /hr) male older than 18 y/o

Exclusion Criteria:

* refuse participate, chronic lung disease active infection neurologic event

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-08; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The levels of IL-6 mRNA expression and activation of NF-B in peripheral blood monocytes were higher in OSA patients than normal subjects. And increased IL-6 mRNA expression and activation of NF-B go down after 4-week CPAP treatment. | patients evaluated before and in the end of four-week after CPAP treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hey-Dong Wu, M.D., Principal Investigator — National Taiwan University Hospital